CLINICAL TRIAL: NCT02226198
Title: A Randomized, Double-blind, Placebo-controlled, Multi-center, Cross-over Study of Rosuvastatin in Children and Adolescents (Aged 6 to <18 Years) With Homozygous Familial Hypercholesterolemia (HoFH)
Brief Title: A Study to Evaluate the Efficacy and Safety of Rosuvastatin in Children and Adolescents With Homozygous Familial Hypercholesterolemia
Acronym: HYDRA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: D3561C00004
Record Dates: First submitted 2014-08-14; First posted 2014-08-27 (Estimated); Results first posted 2016-07-04 (Estimated); Last update posted 2016-07-04 (Estimated); Status verified 2016-07

CONDITIONS: Homozygous Familial Hypercholesterolemia (HoFH)
Keywords: LDL-C; HoFH; Hyperlipidemia
MeSH Terms: conditions — Homozygous Familial Hypercholesterolemia; Hyperlipidemias | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rosuvastatin (Active Comparator): 6-week treatment period, and after crossover finished a 12-week efficacy maintenance phase for all patients
  Interventions: Drug: Rosuvastatin 20mg
- Placebo (Placebo Comparator): 6 weeks treatment during crossover
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rosuvastatin 20mg — Active drug will be taken taken orally, QD, either in the morning or in the evening
  Arms: Rosuvastatin
Drug: Placebo — Will be taken taken orally, QD, either in the morning or in the evening
  Arms: Placebo

SUMMARY:
The purpose of the study is to establish the efficacy, safety and tolerability of rosuvastatin in children and adolescents with homozygous familial hypercholesterolemia.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, multi-center, cross-over study of the efficacy, safety and tolerability rosuvastatin in children and adolescents (aged 6 to <18 years) with homozygous familial hypercholesterolemia (HoFH). The study is designed to assess the efficacy of rosuvastatin 20 mg compared to placebo on lipids, lipoproteins and apolipoproteins in pediatric patients with HoFH. The outcome measures to be assessed include low density lipoprotein cholesterol (LDL-C), high density lipoprotein cholesterol (HDL-C), total cholesterol (TC), triglycerides, non-HDL-C, LDL-C/HDL-C, TC/HDL-C, non-HDL-C/HDL-C, apolipoprotein B (ApoB), apolipoprotein A 1 (ApoA-1) and ApoB/ApoA-1 following 6 weeks of treatment with rosuvastatin 20 mg or placebo. Pharmacokinetic data of the trough plasma exposure of rosuvastatin will also be assessed in these pediatric patients with HoFH.

ELIGIBILITY:
Inclusion Criteria:

1. Prior to any study related procedures being performed, provision of written informed consent from a parent/both parents or guardian and statement of assent from the child or adolescent (if required by Institutional Review Board [IRB] or Independent Ethics Committee [EC] according to local regulations and guidelines). Communication between the Investigator, patient/guardian and child/adolescent to confirm understanding and required compliance with the requirements of the study.
2. Male and female children and adolescents (aged 6 to <18 years) with at least 1 of the following criteria:

   Documentation of genetic testing confirming 2 mutated alleles of the LDL receptor gene locus; and/or

   Documented untreated LDL C >500 mg/dL (12.9 mmol/L) and triglyceride (TG) <300 mg/dL (3.4 mmol/L) and at least 1 of the following criteria:
   1. Tendinous and/or cutaneous xanthoma prior to 10 years of age; or
   2. Documentation of HoFH in both parents by:

      * genetic and/or
      * clinical criteria
3. Negative pregnancy test (b human chorionic gonadotropin analysis) prior to baseline in females of child bearing potential:

   * Female patients of child bearing potential must adhere to a pregnancy prevention method (abstinence, chemical, or mechanical) during the study and 3 months following the last dose.
   * Male patients should refrain from fathering a child (including sperm donation) during the study and up to 3 months following the last dose; and
4. Willing to follow all study procedures including adherence to dietary guidelines, study visits, fasting blood draws, and compliance with study treatment regimens.

Exclusion Criteria

1. History of statin inducted myopathy or serious hypersensitivity reaction to other HMG CoA reductase inhibitors (statins), including rosuvastatin, at Visit 1.
2. Fasting serum glucose of >9.99 mmol/L (180 mg/dL) or glycosylated hemoglobin >9% at Visit 1 or patients with a history of diabetic ketoacidosis within the past year.
3. Uncontrolled hypothyroidism defined as thyroid stimulating hormone (TSH) >1.5 times the upper limit of normal (ULN) at Visit 1 or patients whose thyroid replacement therapy was initiated or modified within the last 3 months prior to Visit 2.
4. Current active liver disease or hepatic dysfunction (except a confirmed diagnosis of Gilbert's disease) as defined as elevations of 1.5 times the upper limit of normal (ULN) for any age in any of the following liver function tests at Visit 1: Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), or bilirubin.
5. Definite or suspected personal history or family history of clinically significant adverse drug reactions (ADRs), or hypersensitivity to drugs with a similar chemical structure to rosuvastatin as well as other statins.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2014-11; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- Research Site, Brussels (Woluwé-St-Lambert), Belgium
- Research Site, Chicoutimi, Quebec, Canada
- Research Site, København Ø, Denmark
- Research Site, Haifa, Israel
- Malaysia (2):
  - Research Site, Kuala Lumpur
  - Research Site, Kubang Kerian
- Netherlands (2):
  - Research Site, Amsterdam
  - Research Site, Goteborg
- Research Site, Taipei, Taiwan

REFERENCES:
- [Derived] Stein EA, Dann EJ, Wiegman A, Skovby F, Gaudet D, Sokal E, Charng MJ, Mohamed M, Luirink I, Raichlen JS, Sunden M, Carlsson SC, Raal FJ, Kastelein JJP. Efficacy of Rosuvastatin in Children With Homozygous Familial Hypercholesterolemia and Association With Underlying Genetic Mutations. J Am Coll Cardiol. 2017 Aug 29;70(9):1162-1170. doi: 10.1016/j.jacc.2017.06.058. PMID 28838366

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty HoFH patients were recruited to 9 centers within 8 countries (Belgium, Canada, Denmark, Israel, Malaysia, Sweden, Taiwan, and The Netherlands) that participated in the study. FSI date: 03-Nov-2014
Pre-assignment Details: 20 enrolled, 3 withdrew consent, 3 did not fulfil eligibility criteria. Among the 14 left, ten went through 4 week lead-in phase and 4 did not.
Groups:
- Overall: Relevant for the lead-in and maintenance phases
- Rosuva First Then Placebo; Placebo First Then Rosuva: Relevant for the cross-over phase
Period: Lead-in Phase
Arm/Group | Overall | Rosuva First Then Placebo | Placebo First Then Rosuva
Started | 11 | 0 | 0
Completed | 10 | 0 | 0
Not Completed | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Period: Cross-Over: First Intervention (6 Weeks)
Arm/Group | Overall | Rosuva First Then Placebo | Placebo First Then Rosuva
Started | 0 | 7 | 7
Completed | 0 | 6 | 7
Not Completed | 0 | 1 | 0
Not completed — No possibility to draw blood | 0 | 1 | 0
Period: Cross-Over: Second Interv. (6 Weeks)
Arm/Group | Overall | Rosuva First Then Placebo | Placebo First Then Rosuva
Started | 0 | 6 | 7
Completed | 0 | 6 | 7
Not Completed | 0 | 0 | 0
Period: Maintenance Phase (12 Weeks)
Arm/Group | Overall | Rosuva First Then Placebo | Placebo First Then Rosuva
Started | 13 | 0 | 0
Completed | 13 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Number of baseline participants are not the same as started as there was a lead-in phase in between and as 6 of the 20 patients starting did not enter the cross-over phase, the beginning of which defines the baseline.
Groups:
- Cross-over: Cross-over phase
Arm/Group | Cross-over
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: Years] | 10.9 (2.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: LDL-Cholesterol (mg/dL)
Description: Change in low density lipoprotein cholesterol (LDL C) following 6 weeks of rosuvastatin 20 mg compared to 6 weeks of placebo treatment
Time Frame: Samples taken on Day 42 (week 6) and on day 84 (week 12)
Population: 6-17 years HoFH
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- C-FAS Rosuvastatin: Cross-over Full Analysys Set, 6 weeks of Rosuvastatin
- C-FAS Placebo: Cross-over Full Analysis Set, 6 weeks of Placebo
Arm/Group | C-FAS Rosuvastatin | C-FAS Placebo
Number analyzed (Participants) | 13 | 13
mg/dL | 396.0 (195.99) | 481.4 (184.90)
Statistical Analysis 1: Comparison: C-FAS Rosuvastatin vs C-FAS Placebo; cross-over, null hypothesis is no difference between ros and plc. Powered for 90% detection of 15% delta; Test type: Superiority or Other; p = 0.005, Mixed Models Analysis — statistical significance set at 0.05; Relative difference in geometric LSM = -22.3, 95% CI 2-sided [-33.5 to -9.1] — Rosuvastatin treatment gives on average a 22.3% lower geometric LS mean than placebo

2. Primary Outcome: LDL-Cholesterol (mmol/L)
Description: as for outcome 1
Time Frame: Samples taken on Day 42 (week 6) and on day 84 (week 12)
Population: 6-17 years HoFH
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | C-FAS Rosuvastatin | C-FAS Placebo
Number analyzed (Participants) | 13 | 13
mmol/L | 10.26 (5.076) | 12.47 (4.790)
Statistical Analysis 1: Comparison: C-FAS Rosuvastatin vs C-FAS Placebo; cross-over, null hypothesis is no difference between ros and plc. Powered for 90% detection of 15% delta; Test type: Superiority or Other; p = 0.005, Mixed Models Analysis — statistical significance set at 0.05; Relative difference in geometric LSM = -22.3, 95% CI 2-sided [-33.5 to -9.1] — Rosuvastatin treatment gives on average a 22.3% lower geometric LS mean than placebo

3. Secondary Outcome: TC (mg/dL)
Description: Efficacy in terms of total cholesterol (TC)
Time Frame: Samples taken at Day 42 (week 6) and Day 84 (week 12)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | C-FAS Rosuvastatin | C-FAS Placebo
Number analyzed (Participants) | 13 | 13
mg/dL | 447.6 (195.46) | 539.0 (184.91)
Statistical Analysis 1: Comparison: C-FAS Rosuvastatin vs C-FAS Placebo; cross-over, null hypothesis is no difference between ros and plc; Test type: Superiority or Other; p = 0.003, Mixed Models Analysis — statistical significance set at 0.05; Relative difference in geometric LSM = -20.1, 95% CI 2-sided [-29.7 to -9.1]

4. Secondary Outcome: TC (mmol/L)
Description: Efficacy in terms of total cholesterol (TC)
Time Frame: Samples taken at Day 42 (week 6) and Day 84 (week 12)
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | C-FAS Rosuvastatin | C-FAS Placebo
Number analyzed (Participants) | 13 | 13
mmol/L | 11.59 (5.063) | 13.96 (4.790)
Statistical Analysis 1: Comparison: C-FAS Rosuvastatin vs C-FAS Placebo; cross-over, null hypothesis is no difference between ros and plc; Test type: Superiority or Other; p = 0.003, Mixed Models Analysis — statistical significance set at 0.05; Relative difference in geometric LSM = -20.1, 95% CI 2-sided [-29.7 to -9.1]

5. Secondary Outcome: Non-HDL C (mg/dL)
Description: Efficacy in terms of non-high density lipoprotein cholesterol (non-HDL C)
Time Frame: Samples taken at Day 42 (week 6) and Day 84 (week 12)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | C-FAS Rosuvastatin | C-FAS Placebo
Number analyzed (Participants) | 13 | 13
mg/dL | 412.1 (198.62) | 505.3 (186.39)
Statistical Analysis 1: Comparison: C-FAS Rosuvastatin vs C-FAS Placebo; cross-over, null hypothesis is no difference between ros and plc; Test type: Superiority or Other; p = 0.003, Mixed Models Analysis — statistical significance set at 0.05; Relative difference in geometric LSM = -22.9, 95% CI 2-sided [-33.7 to -10.3]

6. Secondary Outcome: Non-HDL C (mmol/L)
Description: Efficacy in terms of non-high density lipoprotein cholesterol (non-HDL C)
Time Frame: Samples taken at Day 42 (week 6) and Day 84 (week 12)
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | C-FAS Rosuvastatin | C-FAS Placebo
Number analyzed (Participants) | 13 | 13
mmol/L | 10.67 (5.144) | 13.09 (4.826)
Statistical Analysis 1: Comparison: C-FAS Rosuvastatin vs C-FAS Placebo; cross-over, null hypothesis is no difference between ros and plc; Test type: Superiority or Other; p = 0.003, Mixed Models Analysis — statistical significance set at 0.05; Relative difference in geometric LSM = -22.9, 95% CI 2-sided [-33.7 to -10.3]

7. Secondary Outcome: ApoB (mg/dL)
Description: Efficacy in terms of apolipoprotein B (ApoB)
Time Frame: Samples taken at Day 42 (week 6) and Day 84 (week 12)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | C-FAS Rosuvastatin | C-FAS Placebo
Number analyzed (Participants) | 13 | 13
mg/dL | 234.9 (107.02) | 267.9 (86.33)
Statistical Analysis 1: Comparison: C-FAS Rosuvastatin vs C-FAS Placebo; cross-over, null hypothesis is no difference between ros and plc; Test type: Superiority or Other; p = 0.024, Mixed Models Analysis — statistical significance set at 0.05; Relative difference in geometric LSM = -17.1, 95% CI 2-sided [-29.2 to -2.9]

8. Secondary Outcome: ApoB (g/L)
Description: Efficacy in terms of apolipoprotein B (ApoB)
Time Frame: Samples taken at Day 42 (week 6) and Day 84 (week 12)
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | C-FAS Rosuvastatin | C-FAS Placebo
Number analyzed (Participants) | 13 | 13
g/L | 2.35 (1.070) | 2.68 (0.863)
Statistical Analysis 1: Comparison: C-FAS Rosuvastatin vs C-FAS Placebo; cross-over, null hypothesis is no difference between ros and plc; Test type: Superiority or Other; p = 0.024, Mixed Models Analysis — statistical significance set at 0.05; Relative difference in geometric LSM = -17.1, 95% CI 2-sided [-29.2 to -2.9]

9. Secondary Outcome: HDL-C (mg/dL)
Description: Efficacy in terms of high density lipoprotein cholesterol (HDL C)
Time Frame: Samples taken at Day 42 (week 6) and Day 84 (week 12)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | C-FAS Rosuvastatin | C-FAS Placebo
Number analyzed (Participants) | 13 | 13
mg/dL | 35.5 (7.29) | 33.7 (8.47)
Statistical Analysis 1: Comparison: C-FAS Rosuvastatin vs C-FAS Placebo; cross-over, null hypothesis is no difference between ros and plc; Test type: Superiority or Other; p = 0.314, Mixed Models Analysis — statistical significance set at 0.05; Relative difference in geometric LSM = 7.4, 95% CI 2-sided [-7.4 to 24.5]

10. Secondary Outcome: HDL-C (mmol/L)
Description: Efficacy in terms of high density lipoprotein cholesterol (HDL C)
Time Frame: Samples taken at Day 42 (week 6) and Day 84 (week 12)
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | C-FAS Rosuvastatin | C-FAS Placebo
Number analyzed (Participants) | 13 | 13
mmol/L | 0.92 (0.189) | 0.87 (0.218)
Statistical Analysis 1: Comparison: C-FAS Rosuvastatin vs C-FAS Placebo; cross-over, null hypothesis is no difference between ros and plc; Test type: Superiority or Other; p = 0.314, Mixed Models Analysis — statistical significance set at 0.05; Relative difference in geometric LSM = 7.4, 95% CI 2-sided [-7.4 to 24.5]

11. Secondary Outcome: LDL-C, Not on Apheresis (mg/dL)
Description: Efficacy in terms of low density lipoprotein cholesterol (LDL C) following 6 weeks rosuvastatin 20 mg or placebo treatment in patients not treated with Apheresis
Time Frame: Samples taken at Day 42 (week 6) and Day 84 (week 12)
Population: Patients not treated with apheresis
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | C-FAS Rosuvastatin | C-FAS Placebo
Number analyzed (Participants) | 6 | 6
mg/dL | 479.8 (239.07) | 594.7 (203.60)
Statistical Analysis 1: Comparison: C-FAS Rosuvastatin; cross-over, null hypothesis is no difference between ros and plc; Test type: Superiority or Other; p = 0.080, Mixed Models Analysis — statistical significance set at 0.05; Relative difference in geometric LSM = -26.3, 95% CI 2-sided [-48.7 to 6.0]

12. Secondary Outcome: LDL-C, Not on Apheresis (mmol/L)
Description: as for outcome 11
Time Frame: Samples taken at Day 42 (week 6) and Day 84 (week 12)
Population: Patients not treated with apheresis
Measure: Mean (Standard Deviation); unit: mmol/L
Groups:
- C-FAS Placebo Not on Apheresis: Cross-over Full Analysis Set, 6 weeks of Placebo
Arm/Group | C-FAS Rosuvastatin | C-FAS Placebo Not on Apheresis
Number analyzed (Participants) | 6 | 6
mmol/L | 12.43 (6.191) | 15.40 (5.274)
Statistical Analysis 1: Comparison: C-FAS Rosuvastatin; cross-over, null hypothesis is no difference between ros and plc; Test type: Superiority or Other; p = 0.080, Mixed Models Analysis — statistical significance set at 0.05; Relative difference in geometric LSM = -26.3, 95% CI 2-sided [-48.7 to 6.0]

13. Secondary Outcome: LDL-C From End of Placebo (mg/dL)
Description: Change in low density lipoprotein cholesterol (LDL C) from end of placebo period to 6, 12, and 18 weeks of therapy with rosuvastatin 20 mg
Time Frame: Samples taken at Day 42 (week 6), Day 84 (week 12), Day 126 (week 18) and Day 168 (week 24)
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- M-FAS Rosuvastatin: Maintenance Full Analysis Set, starting cross-over phase with 6 weeks of rosuvastatin
- M-FAS Placebo: Maintenance Full Analysis Set, starting cross-over phase with 6 weeks of placebo
Arm/Group | M-FAS Rosuvastatin | M-FAS Placebo
Number analyzed (Participants) | 7 | 6
mg/dL
  End of Placebo | 472.9 (171.77) | 491.3 (215.46)
  6 weeks after end of Placebo | 399.4 (214.28) | 421.7 (224.49)
  12 weeks after end of Placebo | 345.8 (214.69) | 394.7 (178.45)
  18 weeks after end of Placebo | NA (NA) — No measurements available since taken only at 6 and 12 weeks after end of placebo | 441.8 (260.31)

14. Secondary Outcome: LDL-C From End of Placebo (mmol/L)
Description: as for outcome 13
Time Frame: Samples taken at Day 42 (week 6), Day 84 (week 12), Day 126 (week 18) and Day 168 (week 24)
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | M-FAS Rosuvastatin | M-FAS Placebo
Number analyzed (Participants) | 7 | 6
mmol/L
  End of Placebo | 12.25 (4.449) | 12.73 (5.583)
  6 weeks after end of Placebo | 10.34 (5.551) | 10.92 (5.813)
  12 weeks after end of Placebo | 8.96 (5.558) | 10.22 (4.621)
  18 weeks after end of Placebo | NA (NA) — No measurements available since taken only at 6 and 12 weeks after end of placebo | 11.44 (6.740)

15. Secondary Outcome: Trough Concentrations
Description: Pharmacokinetic profile in terms of trough concentrations. Cross-over phase results based on measurements taken after 6 weeks active treatment (rosuvastatin) in the cross-over phase. Maintenance phase results based on measurements taken after 6 weeks active treatment (rosuvastatin) in the maintenance phase.
Time Frame: Samples taken 24 hours post-dose at Day 42 (week 6), Day 84 (week 12), Day 126 (week 18)
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Cross-over Phase: Measurements taken after 6 weeks active treatment (rosuvastatin) in the cross-over phase
- Maintenance Phase: Measurement taken after 6 weeks active treatment (rosuvastatin) in the maintenance phase.
Arm/Group | Cross-over Phase | Maintenance Phase
Number analyzed (Participants) | 11 | 13
ng/mL | 7.387 (8.11) | 4.482 (3.50)

16. Secondary Outcome: Adverse Events
Description: Safety and tolerability will be described in terms of frequency and severity of adverse events
Time Frame: From screening (5-6weeks before dose) up to the last visit Day 168 (approximately 30 weeks after screening)
Measure: Number; unit: adverse events
Groups:
- Lead-in: Optional 10mg lead-in phase, Safety analysis set
- Cross-over Phase: Cross-over phase, Safety analysis set
- Maintenance: Maintenance Phase, Safety analysis set
Arm/Group | Lead-in | Cross-over Phase | Maintenance
Number analyzed (Participants) | 11 | 14 | 13
adverse events
  Any AE | 4 | 5 | 1
  Any TEAE | 4 | 5 | 1
  Any AE leading to death | 0 | 0 | 0
  Any SAE | 0 | 0 | 0

17. Secondary Outcome: AE's Leading to Discontinuation
Description: Safety and tolerability will be described in terms of rate of discontinuations due to adverse events
Time Frame: From screening (5-6weeks before dose) up to the last visit Day 168 (approximately 30 weeks after screening)
Measure: Number; unit: adverse events
Groups:
- Maintenance Phase: Maintenance phase, Safety analysis set
Arm/Group | Lead-in | Cross-over Phase | Maintenance Phase
Number analyzed (Participants) | 11 | 14 | 13
adverse events | 0 | 0 | 0

18. Secondary Outcome: Abnormal Serum Levels
Description: Safety and tolerability will be described in terms of abnormal serum laboratory values. The reported parameters are not the only ones measured, but rather those for which abnormailities were found
Time Frame: From screening (5-6weeks before dose) up to the last visit Day 168 (approximately 30 weeks after screening)
Measure: Number; unit: participants
Groups:
- Ros/Pla <LLN; Ros/Pla >ULN: Safety Analysis Set, starting cross-over phase with 6 weeks of rosuvastatin
- Pla/Ros <LLN; Pla/Ros >ULN: Safety Analysis Set, starting cross-over phase with 6 weeks of placebo
Arm/Group | Ros/Pla <LLN | Ros/Pla >ULN | Pla/Ros <LLN | Pla/Ros >ULN
Number analyzed (Participants) | 7 | 7 | 7 | 7
participants
  Alanine Aminotransferase week 0 | 0 | 0 | 0 | 0
  Alanine Aminotransferase week 6 | 0 | 1 | 0 | 0
  Alanine Aminotransferase week 12 | 0 | 0 | 0 | 1
  Alanine Aminotransferase week 18 | 0 | 0 | 0 | 1
  Alanine Aminotransferase week 24 | 0 | 1 | 0 | 0
  Albumin week 0 | 0 | 0 | 0 | 1
  Albumin week 6 | 0 | 0 | 0 | 0
  Albumin week 12 | 0 | 0 | 0 | 0
  Albumin week 18 | 0 | 0 | 0 | 1
  Albumin week 24 | 0 | 0 | 0 | 0
  Bicarbonate week 0 | 1 | 0 | 0 | 1
  Bicarbonate week 6 | 0 | 0 | 1 | 0
  Bicarbonate week 12 | 1 | 0 | 1 | 0
  Bicarbonate week 18 | 0 | 0 | 1 | 0
  Bicarbonate week 24 | 1 | 0 | 1 | 0
  Blood Urea Nitrogen week 0 | 1 | 0 | 0 | 0
  Blood Urea Nitrogen week 6 | 1 | 0 | 0 | 0
  Blood Urea Nitrogen week 12 | 1 | 0 | 0 | 0
  Blood Urea Nitrogen week 18 | 1 | 0 | 0 | 0
  Blood Urea Nitrogen week 24 | 0 | 0 | 0 | 0
  Chloride week 0 | 0 | 2 | 0 | 1
  Chloride week 6 | 0 | 0 | 0 | 1
  Chloride week 12 | 0 | 0 | 0 | 0
  Chloride week 18 | 0 | 1 | 0 | 1
  Chloride week 24 | 0 | 0 | 0 | 0
  Creatine Kinase week 0 | 0 | 0 | 0 | 0
  Creatine Kinase week 6 | 0 | 1 | 0 | 0
  Creatine Kinase week 12 | 0 | 0 | 0 | 0
  Creatine Kinase week 18 | 0 | 0 | 0 | 0
  Creatine Kinase week 24 | 0 | 1 | 0 | 0
  Glucose week 0 | 0 | 1 | 0 | 0
  Glucose week 6 | 0 | 0 | 0 | 1
  Glucose week 12 | 0 | 0 | 0 | 0
  Glucose week 18 | 0 | 1 | 0 | 1
  Glucose week 24 | 0 | 0 | 0 | 0
  Potassium week 0 | 0 | 0 | 0 | 1
  Potassium week 6 | 0 | 0 | 0 | 0
  Potassium week 12 | 0 | 0 | 0 | 0
  Potassium week 18 | 0 | 0 | 0 | 0
  Potassium week 24 | 0 | 0 | 0 | 0
  Protein week 0 | 0 | 0 | 0 | 0
  Protein week 6 | 0 | 0 | 0 | 0
  Protein week 12 | 0 | 0 | 0 | 1
  Protein week 18 | 0 | 0 | 0 | 0
  Protein week 24 | 0 | 0 | 0 | 1
  Sodium week 0 | 2 | 0 | 0 | 0
  Sodium week 6 | 1 | 0 | 0 | 0
  Sodium week 12 | 0 | 0 | 0 | 0
  Sodium week 18 | 3 | 0 | 1 | 0
  Sodium week 24 | 0 | 0 | 2 | 0
  Total Bilirubin week 0 | 0 | 0 | 0 | 0
  Total Bilirubin week 6 | 0 | 1 | 0 | 0
  Total Bilirubin week 12 | 0 | 0 | 0 | 0
  Total Bilirubin week 18 | 0 | 0 | 0 | 0
  Total Bilirubin week 24 | 0 | 0 | 0 | 0
  Urate week 0 | 0 | 1 | 0 | 0
  Urate week 6 | 0 | 1 | 0 | 1
  Urate week 12 | 0 | 1 | 0 | 0
  Urate week 18 | 0 | 1 | 0 | 1
  Urate week 24 | 0 | 1 | 0 | 1
  Ery. Mean Corpuscular HGB Concentration week 0 | 2 | 0 | 3 | 0
  Ery. Mean Corpuscular HGB Concentration week 6 | 0 | 0 | 2 | 0
  Ery. Mean Corpuscular HGB Concentration week 12 | 3 | 0 | 2 | 0
  Ery. Mean Corpuscular HGB Concentration week 18 | 1 | 0 | 2 | 0
  Ery. Mean Corpuscular HGB Concentration week 24 | 2 | 0 | 3 | 0
  Ery. Mean Corpuscular Hemoglobin week 0 | 1 | 0 | 3 | 0
  Ery. Mean Corpuscular Hemoglobin week 6 | 1 | 0 | 2 | 0
  Ery. Mean Corpuscular Hemoglobin week 12 | 2 | 0 | 2 | 0
  Ery. Mean Corpuscular Hemoglobin week 18 | 1 | 0 | 2 | 0
  Ery. Mean Corpuscular Hemoglobin week 24 | 1 | 0 | 2 | 0
  Ery. Mean Corpuscular Volume week 0 | 1 | 0 | 2 | 0
  Ery. Mean Corpuscular Volume week 6 | 1 | 0 | 2 | 0
  Ery. Mean Corpuscular Volume week 12 | 1 | 0 | 2 | 0
  Ery. Mean Corpuscular Volume week 18 | 1 | 0 | 2 | 0
  Ery. Mean Corpuscular Volume week 24 | 1 | 0 | 2 | 0
  Erythrocytes week 0 | 1 | 0 | 0 | 1
  Erythrocytes week 6 | 0 | 0 | 0 | 0
  Erythrocytes week 12 | 0 | 0 | 1 | 1
  Erythrocytes week 18 | 0 | 0 | 1 | 0
  Erythrocytes week 24 | 0 | 2 | 0 | 2
  Hematocrit week 0 | 2 | 0 | 2 | 0
  Hematocrit week 6 | 2 | 0 | 3 | 0
  Hematocrit week 12 | 1 | 0 | 2 | 0
  Hematocrit week 18 | 1 | 0 | 3 | 0
  Hematocrit week 24 | 0 | 0 | 1 | 0
  Hemoglobin week 0 | 2 | 0 | 3 | 0
  Hemoglobin week 6 | 2 | 0 | 3 | 0
  Hemoglobin week 12 | 1 | 0 | 3 | 0
  Hemoglobin week 18 | 1 | 0 | 3 | 0
  Hemoglobin week 24 | 0 | 0 | 2 | 0
  Lymphocytes/Leukocytes week 0 | 0 | 0 | 0 | 1
  Lymphocytes/Leukocytes week 6 | 0 | 0 | 0 | 1
  Lymphocytes/Leukocytes week 12 | 0 | 0 | 0 | 1
  Lymphocytes/Leukocytes week 18 | 0 | 1 | 0 | 1
  Lymphocytes/Leukocytes week 24 | 0 | 1 | 0 | 1
  Neutrophils, Segmented/Leukocytes week 0 | 0 | 0 | 0 | 0
  Neutrophils, Segmented/Leukocytes week 6 | 0 | 0 | 0 | 0
  Neutrophils, Segmented/Leukocytes week 12 | 0 | 0 | 0 | 0
  Neutrophils, Segmented/Leukocytes week 18 | 1 | 0 | 0 | 0
  Neutrophils, Segmented/Leukocytes week 24 | 1 | 0 | 0 | 0
  Neutrophils/Leukocytes week 0 | 0 | 0 | 0 | 0
  Neutrophils/Leukocytes week 6 | 1 | 0 | 0 | 0
  Neutrophils/Leukocytes week 12 | 0 | 0 | 0 | 0
  Neutrophils/Leukocytes week 18 | 0 | 0 | 0 | 0
  Neutrophils/Leukocytes week 24 | 0 | 0 | 0 | 0
  Platelets week 0 | 0 | 1 | 0 | 0
  Platelets week 6 | 0 | 0 | 0 | 1
  Platelets week 12 | 0 | 0 | 0 | 0
  Platelets week 18 | 0 | 0 | 0 | 0
  Platelets week 24 | 0 | 0 | 0 | 1

19. Secondary Outcome: Height
Description: Safety and tolerability will be described in terms of growth, including height (linear growth [cm and standard deviation (SD) score]), and weight.
Time Frame: Week 0 (start of cross-over), weeks 6, week 12 and week 18
Measure: Mean (Standard Deviation); unit: cm
Groups:
- Ros/Pla: Safety Analysis Set, starting cross-over with 6 weeks of rosuvastatin
- Pla/Ros: Safety Analysis Set, starting crossover-phase with 6 weeks of placebo
Arm/Group | Ros/Pla | Pla/Ros
Number analyzed (Participants) | 7 | 7
cm
  Height (cm) week 0 | 144.0 (17.82) | 140.9 (15.70)
  Height (cm) week 6 | 144.9 (17.70) | 141.1 (16.11)
  Height (cm) week 12 | 145.7 (18.07) | 142.0 (17.17)
  Height (cm) week 18 | 146.9 (17.68) | 142.3 (16.99)
  Height (cm) week 24 | 147.1 (17.94) | 143.5 (17.58)

20. Secondary Outcome: Height Z-score
Description: as for outcome 19
Time Frame: Week 0 (start of cross-over), weeks 6, week 12 and week 18
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Ros/Pla | Pla/Ros
Number analyzed (Participants) | 7 | 7
ratio
  Height z-score week 0 | -0.42 (1.697) | -0.75 (1.555)
  Height z-score week 6 | -0.29 (1.703) | -0.71 (1.644)
  Height z-score week 12 | -0.18 (1.742) | -0.70 (1.776)
  Height z-score week 18 | 0.00 (1.721) | -0.65 (1.757)
  Height z-score week 24 | 0.04 (1.752) | -0.49 (1.758)

21. Secondary Outcome: Weight
Description: as for outcome 19
Time Frame: Week 0 (start of cross-over), weeks 6, week 12 and week 18
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Ros/Pla | Pla/Ros
Number analyzed (Participants) | 7 | 7
kg
  Weight (kg) week 0 | 37.39 (12.731) | 40.19 (16.520)
  Weight (kg) week 6 | 38.14 (13.577) | 40.36 (16.462)
  Weight (kg) week 12 | 38.63 (14.426) | 42.30 (18.651)
  Weight (kg) week 18 | 39.31 (14.588) | 42.50 (17.990)
  Weight (kg) week 24 | 39.90 (14.550) | 43.00 (17.867)

22. Secondary Outcome: Tanner Stage
Description: Stages for fem (Pubic hair, Breasts):
  1. (Preadol,Preadol)
  2. (Sparse, lightly pigmented, medial border of labia,Breast and papilla elevated as small mound; areolar diam incr)
  3. (Darker, beginning to curl, incr amount, Breast and areola enlarged, no contour separation)
  4. (Course, curly, abundant but less amount in adult,Areola and papilla form secondary mound)
  5. (Adult fem triangle, spread to medial surface of thighs,Mature, nipple projects, areola part of general breast contour) For males (Pubic hair, Penis, Testes)
  1=(None,Preadol,Preadol) 2=(Scanty, long, light pigm,Slight enl,Enl scrotum, pink texture alt) 3=(Darker, starts to curl, small amount,Longer,Larger) 4=(Resembles adult type, but less in quant; course, curly,Larger; glans and breadth increased in size,Larger, scrotum dark) 5=(Adult distr, spread to medial thighs,Adult size,Adult size). Progr at a normal rate is preferred. Regr is not preferred.
Time Frame: Week 0 (start of cross-over)
Measure: Mean (Standard Deviation); unit: stage
Arm/Group | Ros/Pla | Pla/Ros
Number analyzed (Participants) | 7 | 7
stage
  Tanner stage week 0 | 2.0 (1.41) | 1.7 (1.11)
  Tanner stage week 24 | 2.3 (1.38) | 2.0 (0.2)

23. Secondary Outcome: TG (mg/dL)
Description: Efficacy in terms of triglycerides (TG)
Time Frame: Samples taken at Day 42 (week 6) and Day 84 (week 12)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | C-FAS Rosuvastatin | C-FAS Placebo
Number analyzed (Participants) | 13 | 13
mg/dL | 79.8 (24.48) | 119.5 (52.67)
Statistical Analysis 1: Comparison: C-FAS Rosuvastatin vs C-FAS Placebo; cross-over, null hypothesis is no difference between ros and plc; Test type: Superiority or Other; p = 0.004, Mixed Models Analysis — statistical significance set at 0.05; Relative difference in geometric LSM = -30.4, 95% CI 2-sided [-44.2 to -13.3]

24. Secondary Outcome: TG (mmol/L)
Description: Efficacy in terms of triglycerides (TG)
Time Frame: Samples taken at Day 42 (week 6) and Day 84 (week 12)
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | C-FAS Rosuvastatin | C-FAS Placebo
Number analyzed (Participants) | 13 | 13
mmol/L | 0.90 (0.277) | 1.35 (0.595)
Statistical Analysis 1: Comparison: C-FAS Rosuvastatin vs C-FAS Placebo; cross-over, null hypothesis is no difference between ros and plc; Test type: Superiority or Other; p = 0.004, Mixed Models Analysis — statistical significance set at 0.05; Relative difference in geometric LSM = -30.4, 95% CI 2-sided [-44.2 to -13.3]

25. Secondary Outcome: LDL C/HDL C
Description: Efficacy in terms of low density lipoprotein cholesterol (LDL C) / high density lipoprotein cholesterol (HDL C)
Time Frame: Samples taken at Day 42 (week 6) and Day 84 (week 12)
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | C-FAS Rosuvastatin | C-FAS Placebo
Number analyzed (Participants) | 13 | 13
ratio | 12.208 (7.8638) | 15.600 (9.1317)
Statistical Analysis 1: Comparison: C-FAS Rosuvastatin vs C-FAS Placebo; cross-over, null hypothesis is no difference between ros and plc; Test type: Superiority or Other; p = 0.006, Mixed Models Analysis — statistical significance set at 0.05; Relative difference in geometric LSM = -27.6, 95% CI 2-sided [-41.2 to -11.0]

26. Secondary Outcome: TC/HDL C
Description: Efficacy in terms of total cholesterol (TC) / high density lipoprotein cholesterol (HDL C)
Time Frame: Samples taken at Day 42 (week 6) and Day 84 (week 12)
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | C-FAS Rosuvastatin | C-FAS Placebo
Number analyzed (Participants) | 13 | 13
ratio | 13.704 (8.0414) | 17.416 (9.5454)
Statistical Analysis 1: Comparison: C-FAS Rosuvastatin vs C-FAS Placebo; cross-over, null hypothesis is no difference between ros and plc; Test type: Superiority or Other; p = 0.005, Mixed Models Analysis — statistical significance set at 0.05; Relative difference in geometric LSM = -25.6, 95% CI 2-sided [-38.1 to -10.5]

27. Secondary Outcome: Non-HDL C/HDL C
Description: Efficacy in terms of non-high density lipoprotein cholesterol (non-HDL C) / HDL C
Time Frame: Samples taken at Day 42 (week 6) and Day 84 (week 12)
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | C-FAS Rosuvastatin | C-FAS Placebo
Number analyzed (Participants) | 13 | 13
ratio | 12.704 (8.0414) | 16.416 (9.5454)
Statistical Analysis 1: Comparison: C-FAS Rosuvastatin; cross-over, null hypothesis is no difference between ros and plc; Test type: Superiority or Other; p = 0.005, Mixed Models Analysis — statistical significance set at 0.05; Relative difference in geometric LSM = -28.2, 95% CI 2-sided [-41.7 to -11.4]

28. Secondary Outcome: ApoB/ApoA
Description: Efficacy in terms of apolipoprotein B (ApoB) / apolipoprotein A (ApoA)
Time Frame: Samples taken at Day 42 (week 6) and Day 84 (week 12)
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | C-FAS Rosuvastatin | C-FAS Placebo
Number analyzed (Participants) | 13 | 13
ratio | 2.408 (1.3259) | 2.873 (1.4669)
Statistical Analysis 1: Comparison: C-FAS Rosuvastatin; cross-over, null hypothesis is no difference between ros and plc; Test type: Superiority or Other; p = 0.013, Mixed Models Analysis — statistical significance set at 0.05; Relative difference in geometric LSM = -20.4, 95% CI 2-sided [-32.8 to -5.6]

29. Secondary Outcome: Urinalysis Abnormalitites
Description: Safety and tolerability will be described in terms of abnormal urine laboratory values
Time Frame: Week 0, week 6, week 12 and week 18
Measure: Number; unit: participants
Groups:
- Ros/Pla: Safety Analysis Set, starting crossover-phase with 6 weeks of rosuvastatin
Arm/Group | Ros/Pla | Pla/Ros
Number analyzed (Participants) | 7 | 7
participants
  Urine Protein week 0 | 3 | 2
  Urine Protein week 6 | 1 | 2
  Urine Protein week 12 | 3 | 2
  Urine Protein week 18 | 2 | 1
  Urine Protein week 24 | 2 | 1
  Urine Ketones week 0 | 1 | 0
  Urine Ketones week 6 | 0 | 0
  Urine Ketones week 12 | 0 | 0
  Urine Ketones week 18 | 0 | 1
  Urine Ketones week 24 | 0 | 0
  Urine Blood week 0 | 1 | 2
  Urine Blood week 6 | 2 | 1
  Urine Blood week 12 | 1 | 2
  Urine Blood week 18 | 1 | 1
  Urine Blood week 24 | 1 | 1

30. Secondary Outcome: ECG Abnormalities
Description: Safety and tolerability will be described in terms of abnormal electro cardio gram (ECG)
Time Frame: Week 0
Measure: Number; unit: participants
Groups:
- Safety Analysis Set: Safety Analysis Set
Arm/Group | Safety Analysis Set | C-FAS Rosuvastatin | C-FAS Placebo
Number analyzed (Participants) | 14 | 7 | 7
participants | 0 | 0 | 0

31. Secondary Outcome: Physical Exam Abnormalitites
Description: Safety and tolerability will be described in terms of abnormal physical examinations. Only parameters for which abnormalities were found are reported.
Time Frame: Screening, Week 0, week 6, week 12 and week 18, week 24
Measure: Number; unit: participants
Arm/Group | Ros/Pla | Pla/Ros
Number analyzed (Participants) | 7 | 7
participants
  General Appearance screening | 1 | 2
  General Appearance week 0 | 1 | 2
  General Appearance week 6 | 1 | 2
  General Appearance week 12 | 1 | 2
  General Appearance week 18 | 1 | 2
  General Appearance week 24 | 1 | 2
  Head and Neck screening | 0 | 2
  Head and Neck week 0 | 0 | 2
  Head and Neck week 6 | 0 | 2
  Head and Neck week 12 | 0 | 2
  Head and Neck week 18 | 0 | 2
  Head and Neck week 24 | 0 | 1
  Lymph Nodes screening | 0 | 0
  Lymph Nodes week 0 | 0 | 1
  Lymph Nodes week 6 | 0 | 0
  Lymph Nodes week 12 | 0 | 0
  Lymph Nodes week 18 | 0 | 0
  Lymph Nodes week 24 | 0 | 0
  Skin screening | 5 | 2
  Skin week 0 | 5 | 2
  Skin week 6 | 5 | 2
  Skin week 12 | 5 | 2
  Skin week 18 | 5 | 2
  Skin week 24 | 5 | 2

32. Secondary Outcome: Abnormal Vital Signs
Description: Safety and tolerability will be described in terms of abnormal vital signs
Time Frame: From screening (5-6weeks before dose) up to the last visit Day 168 (approximately 30 weeks after screening)
Measure: Number; unit: participants
Arm/Group | Safety Analysis Set
Number analyzed (Participants) | 14
participants | 0

ADVERSE EVENTS:
Groups:
- Lead-in: Lead-in
- Maintenance: Maintenance phase
Arm/Group | Lead-in | Cross-over | Maintenance
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/14 | 0/13
Other Adverse Events (participants affected / at risk) | 4/11 | 4/14 | 1/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lead-in (N=11) | Cross-over (N=14) | Maintenance (N=13)
Influenza like illness (General disorders) | 2 (2) | 2 (2) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Blood bicarbonate decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Upon completion of the Clinical Trial (CT), the Principal Investigator (PI) may prepare the data derived from the CT for publication or presentation. Material should be submitted to the Sponsor for review prior to review or submission for publication, or public dissemination. Publications from individual sites must not precede the primary manuscript, but if not published within twelve months after completion of the CT, the PI has the right to publish or present the methods and results of the CT.